CLINICAL TRIAL: NCT01219621
Title: A Prospective Canadian Multi-Center Randomized Study; Spontaneous AtrioVEntricular Conduction PReservation
Brief Title: Comparison of AAIsafeR and DDD Modes in Non-selected Patients
Acronym: CAN-SAVE R
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorin Group Canada (Industry)
Responsible Party: Bernard Thibault, MD, ICM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGXD04
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2006-09

CONDITIONS: Any Patient Who Fulfills the Inclusion Criteria to be Implanted With a Dual Chamber Pacemaker Maybe Included in the Study as Per ACC/AHA Guidelines
Keywords: Symphony DR 2550,; Dual Chamber Pacemaker,; Sorin,; Ela Medical,; DDD Mode,; AAIsafeR2 mode,; AV-Conduction,; Reducing Ventricular Pacing,; Congestive Heart Failure,; Cardiac Function,; Atrial Arrhythmia,; Atrial Fibrillation,; Atrial and Ventricular Hemodynamics,; Long AV-delays.; Ventricular Function,; Implantation,
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DDD Long AVD (Active Comparator)
  Interventions: Procedure: Symphony Dual Chamber Rate Responsive Device
- safeR (Experimental)
  Interventions: Procedure: Symphony Dual Chamber Rate Responsive Device

INTERVENTIONS:
Procedure: Symphony Dual Chamber Rate Responsive Device — Echocardiography ANP/BNP measurements

SUMMARY:
1 Purpose

In patients with sinus node dysfunction (SND), the use of AAI mode is rare. In paroxysmal high-degree or complete atrio-ventricular (AV) block, paroxysmal vagally-mediated bradycardia, single chamber atrial pacemakers are contraindicated although ventricular support is only rarely needed. As a result, these patients are usually exposed to an unnecessary high proportion of ventricular pacing due to the programming of the system to DDD mode for preventive safety reasons. This drains the pulse generator battery, and more importantly has long-term adverse effects on ventricular function in a subset of vulnerable patients, leading to left ventricular (LV) asynchrony, mitral regurgitation and increased left atrium (LA) size. The deleterious effects of right ventricular (RV) pacing, which increased heart failure (HF) morbidity/mortality, atrial fibrillation (AF) and related adverse events have been highlighted in several large clinical studies. Limiting RV pacing in non-dependant patients is therefore desirable.

The Symphony DR 2550 cardiac pacemakers (SORIN Group, Montrouge, France) offer a new pacing mode that automatically switches from AAI(R) mode to DDD(R) or DDI(R) in event of severe atrioventricular conduction disorder, returning spontaneously to AAI(R) mode as soon as the spontaneous AV conduction has resumed. This particular mode is called the AAIsafeR2(R).

The objective of this study is three-fold: to demonstrate that AAIsafeR2 mode (i) reduces the percentage of ventricular pacing in patients with a spontaneous AV conduction and (ii) prevents atrial arrhythmias by improving atrial hemodynamics and (iii) improves the long-term hemodynamic status of implanted patients in comparison to the "standard" DDD mode, set with long AV Delays (DDD Long AVD).

The scientific soundness lying in this study is a proposal of an optimal programming of dual-chamber pacemakers (PM) with regard to the preservation of spontaneous AV conduction.

DETAILED DESCRIPTION:
In patients with sinus node dysfunction (SND), the use of AAI mode is rare. In paroxysmal high-degree or complete atrio-ventricular (AV) block, paroxysmal vagally-mediated bradycardia, single chamber atrial pacemakers are contraindicated although ventricular support is only rarely needed. As a result, these patients are usually exposed to an unnecessary high proportion of ventricular pacing due to the programming of the system to DDD mode for preventive safety reasons. This drains the pulse generator battery, and more importantly has long-term adverse effects on ventricular function in a subset of vulnerable patients, leading to left ventricular (LV) asynchrony, mitral regurgitation and increased left atrium (LA) size. The deleterious effects of right ventricular (RV) pacing, which increased heart failure (HF) morbidity/mortality, atrial fibrillation (AF) and related adverse events have been highlighted in several large clinical studies. Limiting RV pacing in non-dependant patients is therefore desirable.

The Symphony DR 2550 cardiac pacemakers (SORIN Group, Montrouge, France) offer a new pacing mode that automatically switches from AAI(R) mode to DDD(R) or DDI(R) in event of severe atrioventricular conduction disorder, returning spontaneously to AAI(R) mode as soon as the spontaneous AV conduction has resumed. This particular mode is called the AAIsafeR2(R).

The objective of this study is three-fold: to demonstrate that AAIsafeR2 mode (i) reduces the percentage of ventricular pacing in patients with a spontaneous AV conduction and (ii) prevents atrial arrhythmias by improving atrial hemodynamics and (iii) improves the long-term hemodynamic status of implanted patients in comparison to the "standard" DDD mode, set with long AV Delays (DDD Long AVD).

The scientific soundness lying in this study is a proposal of an optimal programming of dual-chamber pacemakers (PM) with regard to the preservation of spontaneous AV conduction.

2 Study devices

Classification Name Manufacturer Name Cardiovascular permanent pacemaker pulse generator SORIN Group Symphony ™ DR2550

3 Summary of study objectives

The aims of this study are to assess the clinical benefits resulting from AAIsafeR2 by comparison with standard dual chamber programming (DDD) with a long AV Delay.

The benefits will be assessed by comparing the percentage of ventricular pacing, the incidence of atrial arrhythmias, and the evolution of the hemodynamic status as observed through echo parameter and ANP/BNP measurements.

The primary objectives of the study are:

to demonstrate the effectiveness of AAIsafeR2 to preserve natural AV conduction as compared to DDD Long AVD. For this purpose, ventricular pacing ratio as retrieved from PM memory will be assessed on a mid-term period (1 year) by inter-groups comparison of:

* Mean V pacing (%)
* Proportion of patients with a V pacing ratio < 1 %.

to demonstrate the effectiveness of AAIsafeR2 to reduce AF incidence on a long-term basis (3-year follow-up) by analyzing in the randomized branches:

* the cumulative time in AF (as documented by PM memory)
* the total number of AF episodes (as documented by PM memory)
* the number of patients who present a cumulative time in AF>30% of the follow-up period (as documented by PM memory)
* the proportion of patients who turned into persistent AF during the study.
* the proportion of patients who turned into permanent AF during the study.

to compare the effects of AAISafeR2 vs. DDD Long AVD on LV function, mitral regurgitation and LA dimensions on a long-term basis (3-year follow-up) by comparing:

* LV ejection fraction (EF) and volumes
* Left atrium dimensions
* Mitral regurgitation severity as measured by standard echocardiographic methods.

The secondary objectives of this study are to report and compare the following in each randomized arm of the study:

Total mortality CHF-related mortality and hospitalizations Evolution of systemic blood pressures, as estimated by ANP/BNP measurements AF-related adverse events, such as strokes/TIA's and cardioversions The evolution of cardiac asynchrony [inter-ventricular (RV-LV) and intra-ventricular (4 segments), as assessed by TDI technics] The evolution of conduction disturbances in patients presenting unknown or under estimated atrio-ventricular blocks on a long-term basis (intra-group analysis). Stratification by pacing indications and cardiopathies.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria / Indications Any patient who fulfils one or more of the official guidelines to be implanted with a dual-chamber pacemaker (primo-implantation) may be included in the study.

Exclusion Criteria:

Exclusion criteria / Contraindications

The patients presenting with one or more of the following characteristics cannot be included:

* Permanent complete AV block
* Permanent atrial and/or ventricular arrhythmias
* already implanted with a cardioverter-defibrillator (ICD)
* Likely to have a cardiac surgery in the next six months, mainly for:
* severe coronary artery disease
* severe valvular disease
* Refuses to sign an consent form after having received the appropriate information
* Refuses to co-operate
* Not able to understand the study objectives and protocol
* Not available for scheduled follow-up
* With a life expectancy less than one year
* Already included into another clinical study competing with the objectives of the CAN-SAVE R study.
* <18 years old.

Contraindications Any patient to whom a contraindication from device labeling applies shall not be included in the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Percentage of ventricular pacing
Atrial Fibrillation/Atrial Arrhythmia Evolution
Cardiac Function Evolution

SECONDARY OUTCOMES:
Congestive Hear Failure and Atrial Fibrillation Clinical Events
Evolution of conduction Disturbances
Safety Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Thibault, MD, IntMed,Cardiologist, Principal Investigator — Institute de Cardilogie Montreal, Montreal Hear t Institute
Locations (10):
- Canada (10):
  - Grey Nuns hospital, Edmonton, Alberta
  - Royal-Alex hospital, Edmonton, Alberta
  - Kingston General Hospital, Kingston, Ontario
  - Southlake hospital, Newmarket, Ontario
  - St Mike's hospital, Toronto, Ontario
  - Institute de Cardilogie, Montreal Heart Institute, Montreal, Quebec
  - Hotel-Dieu St Jerome, Saint-Jérôme, Quebec
  - Laval hospital, Ste Foy, Quebec
  - Trois-Riviere general hospital, Trois-Rivières, Quebec
  - SASKATOON hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Thibault B, Simpson C, Gagne CE, Blier L, Senaratne M, McNicoll S, Stuglin C, Williams R, Pinter A, Khaykin Y, Nitzsche R. Impact of AV conduction disorders on SafeR mode performance. Pacing Clin Electrophysiol. 2009 Mar;32 Suppl 1:S231-5. doi: 10.1111/j.1540-8159.2008.02293.x. PMID 19250103
- [Derived] Thibault B, Ducharme A, Baranchuk A, Dubuc M, Dyrda K, Guerra PG, Macle L, Mondesert B, Rivard L, Roy D, Talajic M, Andrade J, Nitzsche R, Khairy P; CAN-SAVE R Study Investigators. Very Low Ventricular Pacing Rates Can Be Achieved Safely in a Heterogeneous Pacemaker Population and Provide Clinical Benefits: The CANadian Multi-Centre Randomised Study-Spontaneous AtrioVEntricular Conduction pReservation (CAN-SAVE R) Trial. J Am Heart Assoc. 2015 Jul 23;4(7):e001983. doi: 10.1161/JAHA.115.001983. PMID 26206737